CLINICAL TRIAL: NCT03544242
Title: Nitrite Infusion in Islet Cell Transplantation: Test of Clinical Efficacy and Determination of Cytoprotective Mechanisms
Brief Title: Nitrite Infusion in Islet Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of eligible subjects, lack of staffing
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Blair Smith, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-160901003
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Diabetes
Keywords: Diabetes; Insulin Resistance; Nitrite; Pancreatic islet cells; Autotransplantation; Ischemia reperfusion injury; Mitigation; Cure; Nitric oxide; Sodium nitrite; Islet cell; Survival; Pancreas; Liver
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control group (Active Comparator)
  Interventions: Other: Control
- Pre-Isolation Infusion (Experimental)
  Interventions: Drug: Pre-Isolation Infusion
- Post-Isolation Infusion (Experimental)
  Interventions: Drug: Post-Isolation Infusion

INTERVENTIONS:
Other: Control — A saline infusion will be administered during the pre-isolation and post-isolation phases.
  Arms: Control group
Drug: Pre-Isolation Infusion — A nitrite infusion will be administered during the pre-isolation phase and a saline infusion will be administered during the post-isolation phase.
  Arms: Pre-Isolation Infusion
Drug: Post-Isolation Infusion — A saline infusion will be administered during the pre-isolation phase and a nitrite infusion will be administered during the reperfusion phase.
  Arms: Post-Isolation Infusion

SUMMARY:
This study seeks to investigate the effects of administering nitrite to pancreatic islet cells that have been removed from a patient for autotransplantation.

DETAILED DESCRIPTION:
Patients diagnosed with chronic pancreatitis or recurrent acute pancreatitis may acquire insulin-dependent diabetes due to islet cell destruction. Therefore, islet cell autotransplantation is the optimal therapeutic approach for many of these patients. Islet cell autotransplantation is typically done by excision of the pancreas, followed by isolation of the islet cells and then infusion of these cells into the sinusoids of the liver. Isolation of the islet cells occurs in an ischemic and hypoxic environment, resulting in ischemia reperfusion (IR) injury and destruction of islet cells following infusion into the sinusoids. Hence, strategies to prevent IR injury and subsequent islet cell destruction, such as the administration of inhaled nitric oxide (NO) or sodium nitrite (NaNO2) could enhance islet cell survival following reperfusion, also decreasing long-term insulin requirement. The purpose of this study is to determine if NO administered by infusion in patients undergoing islet cell auto transplantation, will inhibit islet cell destruction, increase diabetes cure rate (decrease the amount of and/or the need for long-term insulin requirement), decrease the ischemic injury (reduces the injury to the islet cells from a decrease in oxygen levels during procurement of the islet cells) during islet cell procurement, and decrease IR injury following islet cell infusion. The primary endpoints of the study are exogenous insulin use, HgbA1c levels post-operatively, and blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age
* Scheduled to undergo Islet Cell auto-transplantation by Dr. Jared White or Dr. Bart Rose
* Subjects who can provide informed written consent and are willing to do so

Exclusion Criteria:

-Any patient with liver disease or unsuitable for surgery (as determined by the surgeon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair Smith, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Started | 1 | 1 | 2
Completed | 1 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion | Total
Number analyzed (Participants) | 1 | 1 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 2 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Prior to Infusion Blood Glucose Serum Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: Between the time of induction and the time immediately prior to infusion of either nitrite or saline
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Pre-islet Cell Infusion Blood Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: Five minutes prior to the infusion of islet cells
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: 20 Minutes After Islet Cells Blood Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 20 minutes after the infusion of Islet Cells
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: 40 Minutes After Islet Cells Blood Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 40 minutes after the infusion of Islet Cells
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: 24 Hours Post Operative Blood Samples Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 24 hours post operatively
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: 48 Hours Post Operative Blood Samples Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 48 hours post operatively
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: 72 Hours Post Operative Blood Samples Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 72 hours post operatively
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: 96 Hours Post Operative Blood Samples Serum Glucose Levels
Description: Blood serum glucose levels will be measured from a blood sample of the amount of 3-5 cc.
Time Frame: 96 hours post operatively
Population: The study did not reach sufficient enrollment power for statistical analysis.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from baseline through 24 months post-operatively
Description: Patients were evaluated for adverse events during appointments.
Arm/Group | Control Group | Pre-Isolation Infusion | Post-Isolation Infusion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03544242/Prot_SAP_000.pdf